CLINICAL TRIAL: NCT01311609
Title: Multi-Site Post Marketing Surveillance Study for Systane in Indian Patients
Brief Title: A Multi-Site Post Marketing Surveillance Study for Systane in Indian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-11-005
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Moderate to Severe Dry Eye
Keywords: Systane, Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane (Experimental): Systane Lubricant Eye Drops
  Interventions: Other: Systane

INTERVENTIONS:
Other: Systane — Systane Lubricant Eye Drops [1-2 Drops in each eye four times daily (QID)]

SUMMARY:
This study is a multi-site, unmasked PMS Study. The purpose of the study is to evaluate the physical effects of Systane Lubricant Eye Drops.

DETAILED DESCRIPTION:
This study is a multi-site, unmasked PMS Study. The purpose of the study is to evaluate the physical effects of Systane Lubricant Eye Drops. The assessed effects include: corneal and conjunctival staining, and ocular signs and symptoms. This is a two week prospective study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, of both sexes, and any race.
* Willing and able to make all required visits and follow study instructions.
* A sodium fluorescein corneal staining sum of >/ 3 in either eye. A best-corrected visual acuity of 0.6 log MAR or better in each eye as assessed during an ETDRS chart

Exclusion Criteria:

* A history or evidence of ocular or intraocular surgery in either eye within the past 6 months.
* Lasik patients can be included if Lasik surgery was > 6 months prior to the initiation of the study.
* A history of intolerance or hypersensitivity to any component of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Corneal Staining | Visit 2 (Week 2) - change from baseline
Best-corrected visual acuity | Visit 2 (Week 2) - change from baseline